CLINICAL TRIAL: NCT05342909
Title: Blood Flow Restriction Training for the Quad: Comparing Daily Training vs. Training Twice a Week
Brief Title: Two Time a Week vs. Five Time a Week Blood Flow Restriction Training Program for the Lower Extremity.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Fox University (Other)
Responsible Party: Principal Investigator, Jason Brumitt, Associate Professor of Physical Therapy, George Fox University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GeorgeFoxU
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Blood Flow Restriction Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5x a week BFR training group (Experimental): Subjects will perform 2 exercises (LAQ and squat) with BFR applied to dominant thigh daily (5x/wk). Exercises performed for 4 sets (30/15/15/15 reps) initially at 30% 1RM; with load increased by 5% every 2 weeks. Training program lasts for 8 weeks. They are also to continue with their regular independent exercise program.
  Interventions: Other: 5x a week BFR training group
- 2x a week BFR training group (Experimental): Subjects will perform 2 exercises (LAQ and squat) with BFR applied to dominant thigh twice a week (2x/wk). Exercises performed for 4 sets (30/15/15/15 reps) initially at 30% 1RM; with load increased by 5% every 2 weeks. Training program lasts for 8 weeks. They are also to continue with their regular independent exercise program.
  Interventions: Other: 2x a week BFR training group
- Control group (No Intervention): This group will not perform any BFR exercises. They are to continue with their regular independent exercise program.

INTERVENTIONS:
Other: 5x a week BFR training group — This group will perform the two exercises 5x a week with blood flow restriction, set to 80% of limb occlusion pressure, applied to the dominant thigh.
  Arms: 5x a week BFR training group
Other: 2x a week BFR training group — This group will perform the two exercises 2x a week with blood flow restriction, set to 80% of limb occlusion pressure, applied to the dominant thigh.
  Arms: 2x a week BFR training group

SUMMARY:
This study will randomize healthy adults who regularly perform resistance training exercises for the lower extremities (2x a week) to one of three groups: a blood flow restriction (BFR) exercise group that trains 2x a week, a BFR exercise group that trains 5x a week, and a control group that does not perform any additional BFR exercise. Those randomized to the BFR groups will perform the unilateral 90-0 knee extension exercise followed by the bilateral squat. Subjects will have the BFR applied to their dominant lower extremity and will perform 4 sets (30/15/15/15 reps) per exercise. Training will initial start at 30% of 1RM with training intensity increased by 5% every 2 weeks. The training program will last 8 weeks.

Pre- and posttests include ultrasound imaging of the dominant leg rectus femoris and strength testing via hand held dynamometry.

ELIGIBILITY:
Inclusion Criteria: healthy adults 18 years of age who currently perform weight-lifting (i.e., resistance training) exercise 2x a week.

-

Exclusion Criteria: current musculoskeletal injury; surgery to the low back or lower extremities during the prior year; one or more contraindications to blood flow restriction training.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Muscular strength | 8 weeks
  Hand held dynamometry will be used to assess changes in strength (bilaterally) for the quadricep, hip extensors, and hip abductors.
Cross-sectional area of the rectus femoris | 8 weeks
  Ultrasound imaging will measure the cross-sectional area of the rectus femoris

CONTACTS AND LOCATIONS:
Overall Officials: JASON BRUMITT, PhD, Principal Investigator — College of Physical Therapy; George Fox University
Locations (2):
- United States (2):
  - George Fox University School of Physical Therapy, Newberg, Oregon
  - George Fox University, Newberg, Oregon

IPD SHARING:
Plan to Share IPD: No